CLINICAL TRIAL: NCT03227133
Title: An Exploratory Study of the Use of Oral Fluency as a Predictive Tool for the Antidepressant Response of Elderly With Unipolar Depressive Disorder
Brief Title: Oral Fluency and the Response to Antidepressant Therapy in the Elderly With a Unipolar Depressive Episode
Acronym: PREDICTage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P/2016/297
Record Dates: First submitted 2017-07-21; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Unipolar Depression
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Psychiatric interview, Neuropsychological evaluations, cardiovascular risk assessment
  Interventions: Other: Neuropsychological evaluations; Other: Psychiatric interview; Other: Cardiovascular risk assessment

INTERVENTIONS:
Other: Neuropsychological evaluations — Neuropsychological evaluations including oral fluency, performed specifically for the study
Other: Psychiatric interview
Other: Cardiovascular risk assessment

SUMMARY:
The study focuses on the identification of clinical, physiological and morphological markers that could predict the response to antidepressant in elderly suffering from unipolar depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Depressive episode according to DSM-5 criteria
* Unipolar depression
* MADRS ≥ 20
* Antidepressive treatment (Serotonin Reuptake Inhibitors/Serotonin Norepinephrine Reuptake Inhibitors)

Exclusion Criteria:

* Other comorbid mental disorders (bipolar disorder, schizophrenia, recent addiction < 3 months except for tobacco)
* Depression with psychotic features
* Serious unstabilized somatic illness
* Protected persons
* Dementia suspected at the time of enrollment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2016-12-23 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06-23 (Estimated)

PRIMARY OUTCOMES:
Ability of the verbal fluency test score to predict the response to antidepressive treatment | week 10
  verbal fluency is assessed during the neuropsychological assessment

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Masse-Sibille, MD, Principal Investigator — Centre Hospitalier Universitaire de Besançon
Locations (1):
- Centre Hospitalier Universitaire de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No